CLINICAL TRIAL: NCT01187719
Title: The Effect of Phenytoin on the Pharmacokinetics of Nevirapine and the Development of Nevirapine Resistance After a Single Dose Nevirapine (VIramune®), Which is Part of ARV Prophylaxis for PMTCT in Moshi, TAnzania, and in Lusaka, Zambia (VITA2 Trial)
Brief Title: The Effect of Phenytoin on the Pharmacokinetics of Nevirapine and the Development of Nevirapine Resistance
Acronym: VITA 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UMCN-AKF 09.02
Record Dates: First submitted 2010-08-23; First posted 2010-08-24 (Estimated); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: HIV-infection; Pregnancy; Mother to Child Transmission
Keywords: HIV; pregnancy; phenytoin; ARV prophylaxis; nevirapine
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Phenytoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): ARV prophylaxis for PMTCT follows national guidelines.
- phenytoin interaction (Experimental): ARV prophylaxis for PMTCT follows national guidelines + start phenytoin 184 mg (2 tablets of 92mg) OD at onset of labour and continue for seven days
  Interventions: Drug: phenytoin

INTERVENTIONS:
Drug: phenytoin — phenytoin 184 mg (2 tablets of 92mg) OD at onset of labour and continue for seven days
  Arms: phenytoin interaction

SUMMARY:
The primary objective of this two-phase trial is as follows:

* To determine the elimination half-life of NVP in HIV positive pregnant women receiving it as a single dose in labour in addition to the ZDV and 3TC with or without seven days phenytoin (pilot PK phase)
* To determine NVP resistance in HIV positive pregnant women receiving it as a single dose in labour in addition to ZDV and 3TC with or without seven days phenytoin (main trial phase)

The secondary objectives of this two-phase trial are as follows:

* To determine the safety of single dose nevirapine with seven days phenytoin as a part of ARV prophylaxis for PMTCT vs. single dose of nevirapine without phenytoin as a part of ARV prophylaxis for PMTCT
* To determine the HIV status of the infant
* To determine the safety of the ARV prophylaxis for PMTCT with seven days of phenytoin on the newborn

Hypothesis: phenytoin reduces the elimination half life of SD NVP and thereby decreases development of resistance to NVP in HIV positive pregnant Tanzanian and Zambian women.

DETAILED DESCRIPTION:
This trial (VITA2) will be done with phenytoin as enzyme inducer to decrease the elimination half-life of NVP as it has also shown a significant difference in the elimination half-life of NVP in the ENVI study and side effects were also transient and mild. The guidelines for ARV prophylaxis for PMTCT has been changed to a more complex regimen. Therefore addition of phenytoin OD for 7 days after delivery will not complicate the regimen for the mother.

Tanzania and Zambia are among the countries in sub-Saharan Africa most affected by the HIV pandemic. In 2008, an estimated 85,000 children were living with HIV in Zambia and out of the 89,000 children born to HIV infected women, 28,000 are infected annually. In Tanzania, 140,000 children were living with HIV in 2007. Both countries use NVP alone or in combination with other drugs as ARV prophylaxis for PMTCT. Little data are available on the extent of NVP resistance in the Tanzanian, Zambian PMTCT setting. Moreover, there is no data available on the follow-up of mother-infant pair with particular focus on resistance to NVP and the infants HIV status. No studies have explored possibilities of reducing NVP resistance by use of an enzyme inducer.

This study seeks to the effect of phenytoin on the pharmacokinetics of NVP and the development of NVP resistance on SD NVP as part of the ARV prophylaxis for PMTCT. This intervention will be part of the VITA2 trial to test the hypothesis that phenytoin reduces the elimination half life of SD NVP and thereby decreases development of resistance to NVP in HIV positive pregnant Tanzanian and Zambian women.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected as documented by positive HIV antibody test
* Antiretroviral naïve
* Starting ARV prophylaxis from 28th weeks of gestation or at least 4 weeks before delivery
* Not intending to relocate out of the area for the duration of study participation
* Willingness of subject to adhere to follow up schedule (note: this is more intensive for the pilot PK phase)
* Ability and willingness of subject to give written consent
* Pregnant women aged 18 years and above
* Willing and able to regularly attend the antenatal clinic

Exclusion Criteria:

* Serious illness that requires systemic treatment or hospitalization
* Use of concomitant medication, which interferes with the ARV prophylaxis for PMTCT or phenytoin
* Any condition that in the opinion of the investigator would compromise the subjects' ability to participate in the study
* Previously treated for HIV infection with antiretroviral agents, including ARV prophylaxis for PMTCT
* Inability to understand the nature and extent of the trial and the procedures required
* CD4 count <350 cells/µl because such a patient is eligible for HAART

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-05; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
half-life time nevirapine | untill two weeks after NVP dosing
  blood samples will be taken <30 min after delivery, 24 hours after delivery, at day 3, at day 5, at day 7 and at day 14

SECONDARY OUTCOMES:
NVP resistance | week 4 / week 6 after delivery
  resistance testing at week 4 or week 6 after delivery (and NVP dosing).
safety of co-administration phenytoin and NVP | entire trial
  Adverse events will be collected during the entire trial (for both mother and child).
HIV status of the newborn | week 6 after birth
  HIV status of the newborn will be assessed at week 6 after birth.

CONTACTS AND LOCATIONS:
Overall Officials: Elton Kisanga, PharmD, PhD, Principal Investigator — Kilimanjaro Christian Medical Centre
Locations (2):
- Kilimanjaro Christian Medical Centre, Moshi, Kilimanjaro, Tanzania
- University Teaching Hospital, Lusaka, Zambia

REFERENCES:
- [Result] Fillekes Q, Muro EP, Chunda C, Aitken S, Kisanga ER, Kankasa C, Thomason MJ, Gibb DM, Walker AS, Burger DM. Effect of 7 days of phenytoin on the pharmacokinetics of and the development of resistance to single-dose nevirapine for perinatal HIV prevention: a randomized pilot trial. J Antimicrob Chemother. 2013 Nov;68(11):2609-15. doi: 10.1093/jac/dkt246. Epub 2013 Jul 17. PMID 23864647